CLINICAL TRIAL: NCT01685294
Title: Effectiveness of Interpersonal Psychotherapy (IPT) for Men and Women Prisoners With Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dr. Jennifer Johnson, Associate Professor (Research), Department of Psychiatry and Human Behavior, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH095230-01 (NIH); R01MH095230 (NIH)
Record Dates: First submitted 2012-08-29; First posted 2012-09-14 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder (MDD); Suicidality; Incarcerated Populations; Prisons; Interpersonal Psychotherapy (IPT)
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (TAU) (No Intervention): Standard prison mental health treatment instead of the research groups, including individual therapy, medication, etc.
- Group Interpersonal Psychotherapy (IPT) for Depression + TAU (Experimental): Participants will receive Group IPT for Depression + TAU.
  Interventions: Behavioral: Group IPT for Depression + TAU

INTERVENTIONS:
Behavioral: Group IPT for Depression + TAU — Interpersonal psychotherapy (IPT) will be administered in 20 group 90-minute sessions over 10 weeks and 4 individual sessions (before group starts, in the middle of the group, at the end of the group, and one month after the group ends). These sessions will focus on improving your relationships with others, building healthy relationships, setting goals, and increasing coping skills. Additionally, participants will receive standard prison mental health treatment, individual therapy, medication, etc.
  Arms: Group Interpersonal Psychotherapy (IPT) for Depression + TAU

SUMMARY:
This study will examine the effects of a first-line treatment for major depressive disorder (MDD), interpersonal psychotherapy (IPT), among men and women prisoners.

DETAILED DESCRIPTION:
The purpose of this 3-year randomized trial is to promote uptake of evidence-based treatment in criminal justice settings by conducting a fully-powered randomized effectiveness study that collects pilot implementation data, including cost-effectiveness data. Group IPT will be compared to treatment as usual (TAU) in a sample of 90 male and 90 female prisoners with MDD from 4 institutions, allowing us to explore gender effects.

ELIGIBILITY:
Inclusion Criteria:

* Meet all DSM-IV criteria for primary (non-substance induced) major depressive disorder
* Expectation of at least 6 months of incarceration at baseline interview
* Incarcerated for at least 4 weeks

Exclusion Criteria:

* Lifetime:

  * Bipolar disorder
  * Psychotic disorder
* Are imminently suicidal
* Cannot understand English well enough to understand the consent form or assessment instruments when read aloud

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2011-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hamilton Rating Scale for Depression (HRSD) at 3 Months | 3 Months from Baseline

SECONDARY OUTCOMES:
Change from Baseline in Suicidality at 3 Months | 3 Months from Baseline
  Suicidality as measured by the Beck Scale for Suicide Ideation.
Change from Baseline in In-Prison Functioning at 3 Months | 3 Months from Baseline
  In-prison functioning will be assessed by the number of correctional programs enrolled/completed and disciplinary/incident reports (measured by the Timeline Followback); aggression/victimization (measured by the Conflict Tactics Scale 2); social support (measured by the Multidimensional Scale of Perceived Social Support and the UCLA Loneliness Scale)
Change from Baseline in Hamilton Rating Scale for Depression (HRSD) at 6 Months | 6 Months from Baseline
Change from Baseline in Suicidality at 6 Months | 6 Months from Baseline
  Suicidality as measured by the Beck Scale for Suicide Ideation.
Change from Baseline in In-Prison Functioning at 6 Months | 6 Months from Baseline
  In-prison functioning will be assessed by the number of correctional programs enrolled/completed and disciplinary/incident reports (measured by the Timeline Followback); aggression/victimization (measured by the Conflict Tactics Scale 2); social support (measured by the Multidimensional Scale of Perceived Social Support and the UCLA Loneliness Scale)
Cost-effectiveness | 6 months post-baseline
  Cost-effectiveness based on costs of IPT and TAU, improvements in HRSD scores, LIFE scores, and cost-offsets, including medical costs, programs completed, fewer fights, fewer suicide attempts, and reduced length of incarceration due to more "good time."

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Johnson, Ph.D., Principal Investigator — Brown University
Locations (5):
- United States (5):
  - Massachusetts Correctional Institute - Old Colony Correctional Center, Bridgewater, Massachusetts
  - Massachusetts Correctional Institution - Framingham, Framingham, Massachusetts
  - South Middlesex Correctional Center, Framingham, Massachusetts
  - Massachusetts Correctional Institution - Norfolk, Norfolk, Massachusetts
  - Adult Correctional Institution - Men's & Women's Medium & Minimum Security Facilities, Cranston, Rhode Island

REFERENCES:
- [Derived] Johnson JE, Hailemariam M, Zlotnick C, Richie F, Wiltsey-Stirman S. Analysis of implementation processes in a hybrid effectiveness-implementation trial of interpersonal psychotherapy (IPT) for major depressive disorder in prisons: Training, supervision, and recommendations. PLoS One. 2024 May 14;19(5):e0288182. doi: 10.1371/journal.pone.0288182. eCollection 2024. PMID 38743716
- [Derived] Felton JW, Hailemariam M, Richie F, Reddy MK, Edukere S, Zlotnick C, Johnson JE. Preliminary efficacy and mediators of interpersonal psychotherapy for reducing posttraumatic stress symptoms in an incarcerated population. Psychother Res. 2020 Feb;30(2):239-250. doi: 10.1080/10503307.2019.1587192. Epub 2019 Mar 11. PMID 30857489
- [Derived] Johnson JE, Stout RL, Miller TR, Zlotnick C, Cerbo LA, Andrade JT, Nargiso J, Bonner J, Wiltsey-Stirman S. Randomized cost-effectiveness trial of group interpersonal psychotherapy (IPT) for prisoners with major depression. J Consult Clin Psychol. 2019 Apr;87(4):392-406. doi: 10.1037/ccp0000379. Epub 2019 Feb 4. PMID 30714749